CLINICAL TRIAL: NCT04919057
Title: Robotic Radical Perineal Prostatectomy for Localized Prostate Cancer: A Feasibility Study
Brief Title: Robotic Radical Perineal Prostatectomy Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chi Hang Yee, Consultant, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRE 2020.019
Record Dates: First submitted 2020-03-23; First posted 2021-06-09 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Robotic Radical Perineal Prostatectomy
Keywords: Robotic Radical Prostatectomy; Perineal; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Robotic perineal radical prostatectomy (Experimental): The patient is laid in the exaggerated lithotomy and 15 degree Trendelenburg position. An incision is made between both ischial tuberosities. Perineal dissection is performed till the apex of the prostate is seen. Subcutaneous tissue laying under the incision borders is dissected deeply over the superficial perineal fascia to place the GelPOINT®.Once the robotic system is docked, dissection of prostate is started.
  Interventions: Device: GelPOINT®

INTERVENTIONS:
Device: GelPOINT® — The patient is laid in the exaggerated lithotomy and 15 degree Trendelenburg position. An incision is made between both ischial tuberosities. Perineal dissection is performed till the apex of the prostate is seen. Subcutaneous tissue laying under the incision borders is dissected deeply over the superficial perineal fascia to place the GelPOINT®.Once the robotic system is docked, dissection of prostate is started.

SUMMARY:
Radical perineal prostatectomy (RPP) was the first approach utilized for the removal of the entire prostate gland for prostate cancer. In the minimally invasive surgery era, the robotic-assisted laparoscopic prostatectomy (RALP) was first described in the early 2000s, and has become the mainstay of prostatectomy in Hong Kong and many parts of the world. Incorporating the robotic technology into the technique of RPP has been studied recently. Some preliminary data showed that such approach resulted in a better functional outcome in continence and erectile function. Our study aims at assessing the safety and effectiveness of robotic RPP in prostate cancer management.

DETAILED DESCRIPTION:
Radical perineal prostatectomy (RPP) was the first approach utilized for the removal of the entire prostate gland for prostate cancer [1]. It continued to be the favoured approach for radical prostatectomy for several decades before the description of the radical retropubic prostatectomy (RRP) by Walsh in 1970s, who has refined the anatomical retropubic approach [2]. In the minimally invasive surgery era, the robotic-assisted laparoscopic prostatectomy (RALP) was first described in the early 2000s [3]. With time, the robotic retropubic approach became one of the most common approaches for prostate removal in prostate cancer patients. In parallel with the implementation of robotic surgery in retropubic prostatectomy, a revival in interest was experienced for the RPP approach in its role for the management of localized prostate cancer. In 2003, Resnick reported a cohort of RPP with reasonable operative times and cancer control concluding that the procedure was safe and effective [4]. Janoff and Parra noted that in comparison to RRP, patients undergoing RPP had less postoperative discomfort, shorter return of bowel function and hospital stay with a decreased transfusion rate [5]. Incorporating the robotic technology into the technique of RPP, Kaouk et al. performed robotic RPP in four patients with localized prostate cancer using a multi-arm da Vinci Surgical system (Intuitive Surgical Inc., Sunnyvale, CA). The procedures were successfully completed applying a robotic perineal approach with patients discharged within 48 hours [6]. Tugku et al reported their clinical experience with 15 patients who underwent robotic RPP [7]. Early continence rate was shown to be 40% at urethral catheter removal and 94% at third months postoperatively. Furthermore, a study was performed by the same group comparing outcomes of robotic RPP versus transperitoneal RALP [8]. Eighty patients (40 robotic RPP vs 40 RALP) with localized prostate cancer were included in the study. Continence rates were 94% in the robotic RPP and 72% in the RALP (p = 0.001) group at the 6th-month follow-up. In terms of erectile function, the rates favoured robotic RPP at 3, 6, and 9-month follow-ups with 44%, 66%, and 75%, respectively. In addition, compared with conventional RALP, robotic RPP would offer an advantage for those patients who had previous intra-abdominal surgery. Moreover, not having the need of putting the patients into steep Trendelenburg position is another potential benefit of robotic RPP over conventional RALP. In this study, we evaluate the early oncological outcome and objective functional outcome of patients undergoing robotic RPP for the treatment of localized prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Men aged between 40 - 80 years
* Localized prostate cancer without obvious lymph node or distant metastases

Exclusion Criteria:

* Clinical T stage T3 or above
* Prostate size >80 ml
* Patients with previous treatment of prostate cancer
* Patients with previous surgery on the prostate
* Patients with active urinary tract infection
* Patients with bladder pathology including bladder stone and bladder cancer
* Patients with urethral stricture
* Patients with neurogenic bladder and/or sphincter abnormalities
* Patients who fail to give informed consent

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only man will develop prostate cancer
Enrollment: 15 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of robotic RPP | During the 1-year post-operation study period
  As defined by completion of prostatectomy via robotic perineal approach

SECONDARY OUTCOMES:
Complications after study intervention | During the 1-year post-operation study period
  Post treatment complication
Positive margin rate | At week-6
  Positive margin rate in the prostatectomy specimen pathology
Disease recurrence | During the 1-year post-operation study period
  Any biochemical recurrence
Functional outcome after robotic RPP | At immediate post-operation, 2-month, 6-month, 9-month and 12-month
  Change in scores in EPIC-26 questionnaires
Quality of life after robotic RRP | At immediate post-operation, 2-month, 6-month, 9-month and 12-month
  Change in scores in IPSS questionnaires

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Davis WH, Scardino PL, Carlton FE. Radical perineal prostatectomy: a 20-year overview. J Urol. 1972 Oct;108(4):604-8. doi: 10.1016/s0022-5347(17)60814-0. No abstract available. PMID 4651353
- [Background] Walsh PC, Lepor H, Eggleston JC. Radical prostatectomy with preservation of sexual function: anatomical and pathological considerations. Prostate. 1983;4(5):473-85. doi: 10.1002/pros.2990040506. PMID 6889192
- [Background] Binder J, Kramer W. Robotically-assisted laparoscopic radical prostatectomy. BJU Int. 2001 Mar;87(4):408-10. doi: 10.1046/j.1464-410x.2001.00115.x. No abstract available. PMID 11251539
- [Background] Resnick MI. Radical perineal prostatectomy. BJU Int. 2003 Oct;92(6):522-3. doi: 10.1046/j.1464-410x.2003.04423.x. No abstract available. PMID 14511023
- [Background] Janoff DM, Parra RO. Contemporary appraisal of radical perineal prostatectomy. J Urol. 2005 Jun;173(6):1863-70. doi: 10.1097/01.ju.0000161483.65619.b3. PMID 15879765
- [Background] Kaouk JH, Akca O, Zargar H, Caputo P, Ramirez D, Andrade H, Albayrak S, Laydner H, Angermeier K. Descriptive Technique and Initial Results for Robotic Radical Perineal Prostatectomy. Urology. 2016 Aug;94:129-38. doi: 10.1016/j.urology.2016.02.063. Epub 2016 May 24. PMID 27233935
- [Background] Tugcu V, Akca O, Simsek A, Yigitbasi I, Sahin S, Tasci AI. Robot-assisted radical perineal prostatectomy: first experience of 15 cases. Turk J Urol. 2017 Dec;43(4):476-483. doi: 10.5152/tud.2017.35488. Epub 2017 Dec 1. PMID 29201511
- [Background] Tugcu V, Akca O, Simsek A, Yigitbasi I, Sahin S, Yenice MG, Tasci AI. Robotic-assisted perineal versus transperitoneal radical prostatectomy: A matched-pair analysis. Turk J Urol. 2019 Apr 3;45(4):265-272. doi: 10.5152/tud.2019.98254. Print 2019 Jul. PMID 30978167
- [Background] Tugcu V, Akca O, Simsek A, Yigitbasi I, Yenice MG, Sahin S, Tasci AI. Robotic perineal radical prostatectomy and robotic pelvic lymph node dissection via a perineal approach: The Tugcu Bakirkoy Technique. Turk J Urol. 2018 Mar;44(2):114-118. doi: 10.5152/tud.2018.24603. Epub 2018 Mar 1. PMID 29511579